CLINICAL TRIAL: NCT05895396
Title: Comparison of Clinical Outcome After Implantation With Two Different Multifocal Toric Intraocular Lens: Liberty Trifocal 677MTY (Medicontur) and PanOptix® Multifocal Toric (Alcon) Lens, With Respect to Rotational Stability, Visual Outcomes, Patients' Satisfaction, YAG Capsulotomy Rate
Brief Title: Clinical Outcome After Implantation of Two Different Multifocal Toric IOLs: Liberty (677MTY) and PanOptix®
Status: Completed | Type: Observational
Sponsor: Medicontur Medical Engineering Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 677MTY _PanOptix_HU_2020
Record Dates: First submitted 2020-12-17; First posted 2023-06-08 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Liberty: The group implanted with Liberty 677MTY
- PanOptix: The group implanted with PanOptix

SUMMARY:
This study is to compare the rotational stability, visual outcome and patient satisfaction after implantation with either Liberty 677MTY, a multifocal diffractive-refractive IOL based on EPS technology manufactured by Medicontur Ltd. (Zsámbék, Hungary) or the multifocal toric IOL PanOptix®, manufactured by Alcon.

DETAILED DESCRIPTION:
According to numerous estimations, 15% to 29% of patients with cataract have more than 1.5 diopters of refractive astigmatism. Corneal astigmatism can be reduced with a variety of surgical techniques including selective positioning of the phacoemulsification incision, corneal relaxing incision, implantation of toric IOLs, photorefractive keratectomy and there are first results of implantation of short arc-length intrastromal corneal ring segments for correcting astigmatism and myopia . The use of toric IOLs to reduce visually significant keratometric astigmatism offers a rational, more predictable and stable method of refractive correction. Implanting a toric intraocular lens offers the possibility of correcting not only spherical equivalent of refraction, but also astigmatism. The success of a toric IOL can be judged not only by its ability to reduce refractive astigmatism immediately postoperatively, but also by its ability to maintain a stable position in the capsular bag in the longer term. Even a small rotational deviation of the toric IOL from its intended axis can result in large reduction of the astigmatic correction.

The purpose of this study is to evaluate and compare the visual outcomes, spectacle independency, visual disturbances (glares, halos), neuronal adaptation and patient satisfaction after implantation of either the Liberty 677MTY (a multifocal diffractive apodized toric intraocular lens- diffractive-refractive IOL based on EPS technology manufactured by Medicontur Ltd. Zsámbék, Hungary) or the multifocal toric PanOptix® IOL, manufactured by Alcon.

ELIGIBILITY:
Inclusion Criteria:

The enrolled subjects will be the patients with cataract and pre-existing regular corneal astigmatism between 1.0 to 6.0 dpt.

Exclusion Criteria:

* astigmatism less than 1 dpt
* irregular astigmatism
* diabetic retinopathy
* iris neovascularisation
* serious intraoperative complications
* congenital eye abnormality
* glaucoma
* pseudoexfoliation syndrom
* amblyopia
* uveitis
* long-term anti-inflammatory treatment
* AMD (advanced AMD)
* retinal detachment
* prior ocular surgery in personal medical history
* corneal diseases
* severe retinal diseases (dystrophy, degeneration)
* severe myopia (if required IOL power is lower than 10 D)
* inadequate visualization of the fundus on preoperative examination
* patients deemed by the clinical investigator because of any systemic disease.
* eye trauma in medical history intraoperative exclusions:
* tear in capsulorhexis
* zonular dehiscence
* posterior capsular rupture
* vitreous loss and other unexpected surgical complication

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with cataract
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Rotational stability | Day 1
  Rotational stability will be measured using slit lamp images of the implanted lens
Rotational stability | 3 months
  Rotational stability will be measured using slit lamp images of the implanted lens
Rotational stability | 1 year
  Rotational stability will be measured using slit lamp images of the implanted lens

SECONDARY OUTCOMES:
Visual outcome (UDVA, CDVA, UIVA, DCIVA, UNVA, DCNVA) | 1 month
  Monocular and binocular visual aquity will be measured at far, intermediate and near by standard ETDRS chart.
Visual outcome (UDVA, CDVA, UIVA, DCIVA, UNVA, DCNVA) | 3 months
  Monocular and binocular visual aquity will be measured at far, intermediate and near by standard ETDRS chart
Visual outcome (UDVA, CDVA, UIVA, DCIVA, UNVA, DCNVA) | 1 year
  Monocular and binocular visual aquity will be measured at far, intermediate and near distances by standard ETDRS chart
Contrast sensitivity defocus curve | 3 months
  Contrast sensitivity defocus curve will be assessed using the Multifocal Lense Analyser iPAD application.
Contrast sensitivity defocus curve | 1 year
  Contrast sensitivity defocus curve will be assessed using the Multifocal Lense Analyser iPAD application.
Contrast sensitivity | 1 year
  Contrast sensitivity in photopic and mesopic light conditions with or without glare will be assessed one year postoperatively using CSV-1000
Multifocality (Visual Acuity Defocus Curve) | 3 months
  The multifocality of the lens will be evaluated also by monocular and binocular visual acuity defocus curves (VADC) using the multifocal lens analyser iPAD application
Multifocality (Visual Acuity Defocus Curve) | 1 year
  The multifocality of the lens will be evaluated also by monocular and binocular visual acuity defocus curves using the multifocal lens analyser iPAD application.
Patient satisfaction | 3 months
  Patient satisfaction will be measures with the VFQ-14 questionnaire
Patient satisfaction | 1 year
  Patient satisfaction will be measures with the VFQ-14 questionnaire

OTHER OUTCOMES:
Safety outcome - Intraoperative complications | Day1 postoperatively
  Intraoperative complications of cataract surgery
  * Posterior capsular or zonular rupture
  * Vitreous loss/anterior vitrectomy or aspiration
  * Iris/ciliary body injury
  * Loss of nuclear material into vitreous
  * Suprachoroidal haemorrhage
  * Retrobulbar haemorrhage
Safety outcome - Postoperative complications | Month1 postoperatively
  Postoperative complications of cataract surgery
  * Cystoid macular oedema
  * Iris abnormalities
  * Corneal oedema
  * Wound leak or rupture
  * IOL dislocation, removal, or exchange
  * Inflammation (Endophthalmitis, anterior chamber cells, anterior chamber flare, hypopyon)
  * Retinal tear, break, or detachment
  * Persistent iritis
  * Elevated intraocular pressure
  * Pupillary block
  * Cornea status
Safety outcome - Complications of IOL implantation | Month 12 postoperatively
  Complications of IOL implantation
  * Posterior capsular opacification (PCO)
  * Opacification, IOL discoloration

CONTACTS AND LOCATIONS:
Overall Officials: József F Győry, MD, Principal Investigator — Retinaszerviz Kft. (8200 Veszprém, Vörösmarty tér 6, Hungary)
Locations (1):
- Retinaszervíz, Veszprém, Hungary